CLINICAL TRIAL: NCT03107611
Title: A Randomized, Prospective, Multicenter, Double Blind, Parallel Assignment, Placebo Controlled Bioequivalence Study of Pimecrolimus Cream, 1% and Elidel® (Pimecrolimus) Cream, 1% in Patients With Mild to Moderate Atopic Dermatitis
Brief Title: Bioequivalence Study of Pimecrolimus Cream, 1% and Elidel® Cream, 1% in Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: DPT Laboratories, Ltd. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CD-14-875
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Results first posted 2020-03-17 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Test (Experimental): Pimecrolimus Cream, 1%, topical, thin layer applied to all affected skin areas twice daily for 14 days
  Interventions: Drug: Pimecrolimus Cream, 1%
- Reference Standard (Active Comparator): Pimecrolimus Cream, 1%, topical, thin layer applied to all affected skin areas twice daily for 14 days
  Interventions: Drug: Pimecrolimus Cream, 1%
- Placebo (Placebo Comparator): Placebo cream, topical, thin layer applied to all affected skin areas twice daily for 14 days
  Interventions: Drug: Placebo Cream

INTERVENTIONS:
Drug: Pimecrolimus Cream, 1%
  Arms: Test
Drug: Placebo Cream
  Arms: Placebo
Drug: Pimecrolimus Cream, 1%
  Other Names: Elidel (pimecrolimus) Cream, 1%
  Arms: Reference Standard

SUMMARY:
To establish the bioequivalence between test drug, Pimecrolimus Cream, 1% with that of reference listed drug, Elidel® (pimecrolimus) Cream 1%, in the treatment of mild to moderate Atopic Dermatitis.

To establish superiority of each active treatment over the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Non-immuno compromised male or female aged 8 years and older
* Clinical diagnosis of mild to moderate Atopic Dermatitis (AD)
* Failed to respond adequately to other topical prescription treatments for AD, or for whom those treatments are not advisable.
* A diagnosis of AD for at least 3 months
* An Investigator's Global Assessment (IGA) of disease severity of mild or moderate at baseline (score of 2 or 3)
* Affected area of AD involvement at least 5% body surface area (BSA)
* Treated with a bland emollient for at least 7 days

Exclusion Criteria:

* Females who are pregnant, breast feeding, or who wish to become pregnant during the study period
* Active cutaneous bacterial or viral infection in any treatment area at baseline (e.g., clinically infected atopic dermatitis, impetigo).
* Sunburn, extensive scarring or pigmented lesion(s) in any treatment area at baseline, which would interfere with evaluations
* History or presence of confounding skin conditions, e.g., psoriasis, rosacea, erythroderma, ichthyosis, or scabies.
* History or presence of Netherton's Syndrome, immunological deficiencies or diseases, HIV, diabetes, malignancy, serious active or recurrent infection, clinically significant severe renal insufficiency or severe hepatic disorders
* Concurrent disease or treatment likely to interfere with the study treatment or evaluations
* Known allergy or hypersensitivity to pimecrolimus or any other component of the drug products
* Not willing to minimize or avoid natural and artificial sunlight exposure during treatment

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (25):
  - Research Facility 6, Boynton Beach, Florida
  - Research Facility 4, Coral Gables, Florida
  - Research Facility 5, Miami, Florida
  - Research Facility 10, Miami, Florida
  - Research Facility 1, Miami Lakes, Florida
  - Research Facility 9, Miramar, Florida
  - Research Facility 33, Sweetwater, Florida
  - Research Facility 23, Boise, Idaho
  - Research Facility 28, Overland Park, Kansas
  - Research Facility 32, Louisville, Kentucky
  - Research Facility 13, New Orleans, Louisiana
  - Research Facility 7, Saint Joseph, Missouri
  - Research Facility 19, Omaha, Nebraska
  - Research Facility 29, Albuquerque, New Mexico
  - Research Facility 24, Charlotte, North Carolina
  - Research Facility 2, High Point, North Carolina
  - Resarch Facility 8, Philadelphia, Pennsylvania
  - Research Facility 18, Johnston, Rhode Island
  - Research Facility 20, Austin, Texas
  - Research Facility 16, College Station, Texas
  - Research Facility 31, Pflugerville, Texas
  - Research Facility 17, Sugar Land, Texas
  - Research Facility 22, West Jordan, Utah
  - Research Facility 15, Richmond, Virginia
  - Research Facility 26, Spokane, Washington
- Research Facility 11, Santo Domingo, Dominican Republic
- Research Facility 12, San Pedro Sula, Honduras

RESULTS

PARTICIPANT FLOW:
Groups:
- Test; Reference Standard: Pimecrolimus Cream, 1%, topical, thin layer applied to all affected skin areas twice daily for 14 days
  Pimecrolimus Cream, 1%
- Placebo: Placebo cream, topical, thin layer applied to all affected skin areas twice daily for 14 days
  Placebo Cream
Period: Overall Study
Arm/Group | Test | Reference Standard | Placebo
Started | 217 | 216 | 221
Dosed (2 Test, 2 Reference, and 1 Placebo Subjects are not known to have dosed) | 215 | 214 | 220
Completed | 210 | 212 | 212
Not Completed | 7 | 4 | 9
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Lost to Follow-up | 3 | 3 | 3
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Worsening signs/symptoms | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Reference Standard | Placebo | Total
Number analyzed (Participants) | 215 | 214 | 220 | 649
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (20.2) | 34.2 (18.9) | 34.9 (21.6) | 35.4 (20.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 144 | 133 | 404
  Male | 88 | 70 | 87 | 245
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 127 | 126 | 125 | 378
  Not Hispanic or Latino | 88 | 88 | 95 | 271
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 3 | 5
  Black or African American | 98 | 93 | 93 | 284
  White | 115 | 118 | 117 | 350
  More than one race | 1 | 1 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 1 | 1
Investigator's Global Assessement of Severity [Count of Participants; unit: Participants]
  Mild | 90 | 96 | 109 | 295
  Moderate | 125 | 118 | 111 | 354

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Modified Intent to Treat Subjects With Success on Investigator's Global Assessment of Disease Severity (Success Being a Score of Clear [0] or Almost Clear [1])
Description: Investigator's Global Assessment of Disease Severity Scale: Clear (0) Minor residual discoloration, no erythema or induration/papulation, no oozing/crusting; Almost Clear (1) Trace faint pink erythema with almost no induration/papulation and no oozing/crusting; Mild disease (1) Faint pink erythema with mild induration/papulation and no oozing/crusting; Moderate disease (3) Pink-red erythema with moderate induration/papulation and there may be some oozing/crusting; Severe disease (4) Deep/bright red erythema with severe induration/papulation with oozing/crusting
Time Frame: Day 15
Population: Modified ITT (Intent-to-treat) sample
Measure: Count of Participants; unit: Participants
Arm/Group | Test | Reference Standard | Placebo
Number analyzed (Participants) | 212 | 212 | 215
Participants | 108 | 115 | 98
Statistical Analysis 1: Comparison: Reference Standard vs Placebo; Test type: Superiority; p = 0.0817, Fisher Exact
Statistical Analysis 2: Comparison: Test vs Placebo; Test type: Superiority; p = 0.2874, Fisher Exact

2. Primary Outcome: Proportion of Per Protocol Subjects With Success on Investigator's Global Assessment of Disease Severity (Success Being a Score of Clear [0] or Almost Clear [1])
Description: as for outcome 1
Time Frame: Day 15
Population: PP (per protocol) sample
Measure: Count of Participants; unit: Participants
Arm/Group | Test | Reference Standard | Placebo
Number analyzed (Participants) | 201 | 205 | 203
Participants | 105 | 113 | 95
Statistical Analysis 1: Comparison: Test vs Reference Standard; Test type: Equivalence — Equivalence margin: -0.20, +0.20; Difference in proportions = -0.03, 90% CI 2-sided [-0.12 to 0.06]

3. Secondary Outcome: Change in Severity of Four Individual Signs and Symptoms
Description: Erythema, induration/papulation, lichenification and pruritus
Time Frame: Day 15
Population: PP sample
Measure: Count of Participants; unit: Participants
Arm/Group | Test | Reference Standard | Placebo
Number analyzed (Participants) | 201 | 205 | 203
Participants
  Erythema - Head & Neck: 3 = Worsen by 3 | 0 | 0 | 0
  Erythema - Head & Neck: 2 = Worsen by 2 | 1 | 1 | 1
  Erythema - Head & Neck: 1 = Worsen by 1 | 2 | 5 | 4
  Erythema - Head & Neck: 0 = No change | 121 | 118 | 135
  Erythema - Head & Neck: -1 = Improve by 1 | 51 | 50 | 48
  Erythema - Head & Neck: -2 = Improve by 2 | 24 | 30 | 15
  Erythema - Head & Neck: -3 = Improve by 3 | 2 | 1 | 0
  Erythema - Trunk: 3 = Worsen by 3 | 0 | 0 | 0
  Erythema - Trunk: 2 = Worsen by 2 | 0 | 1 | 0
  Erythema - Trunk: 1 = Worsen by 1 | 3 | 4 | 6
  Erythema - Trunk: 0 = No change | 106 | 113 | 116
  Erythema - Trunk: -1 = Improve by 1 | 56 | 57 | 50
  Erythema - Trunk: -2 = Improve by 2 | 35 | 30 | 30
  Erythema - Trunk: -3 = Improve by 3 | 1 | 0 | 1
  Erythema - Upper Limbs: 3 = Worsen by 3 | 0 | 0 | 0
  Erythema - Upper Limbs: 2 = Worsen by 2 | 0 | 0 | 1
  Erythema - Upper Limbs: 1 = Worsen by 1 | 4 | 1 | 7
  Erythema - Upper Limbs: 0 = No change | 71 | 80 | 85
  Erythema - Upper Limbs: -1 = Improve by 1 | 76 | 91 | 76
  Erythema - Upper Limbs: -2 = Improve by 2 | 49 | 33 | 33
  Erythema - Upper Limbs: -3 = Improve by 3 | 1 | 0 | 1
  Erythema - Lower Limbs: 3 = Worsen by 3 | 0 | 0 | 0
  Erythema - Lower Limbs: 2 = Worsen by 2 | 0 | 0 | 1
  Erythema - Lower Limbs: 1 = Worsen by 1 | 2 | 4 | 4
  Erythema - Lower Limbs: 0 = No change | 101 | 109 | 106
  Erythema - Lower Limbs: -1 = Improve by 1 | 64 | 62 | 61
  Erythema - Lower Limbs: -2 = Improve by 2 | 34 | 30 | 30
  Erythema - Lower Limbs: -3 = Improve by 3 | 0 | 0 | 1
  Induration/Papulation - Head & Neck: 3 = Worsen by 3 | 0 | 0 | 0
  Induration/Papulation - Head & Neck: 2 = Worsen by 2 | 1 | 2 | 0
  Induration/Papulation - Head & Neck: 1 = Worsen by 1 | 0 | 5 | 3
  Induration/Papulation - Head & Neck: 0 = No change | 118 | 117 | 135
  Induration/Papulation - Head & Neck: -1 = Improve by 1 | 59 | 57 | 51
  Induration/Papulation - Head & Neck: -2 = Improve by 2 | 22 | 23 | 14
  Induration/Papulation - Head & Neck: -3 = Improve by 3 | 1 | 1 | 0
  Induration/Papulation - Trunk: 3 = Worsen by 3 | 0 | 0 | 0
  Induration/Papulation - Trunk: 2 = Worsen by 2 | 0 | 1 | 1
  Induration/Papulation - Trunk: 1 = Worsen by 1 | 5 | 4 | 5
  Induration/Papulation - Trunk: 0 = No change | 103 | 110 | 108
  Induration/Papulation - Trunk: -1 = Improve by 1 | 62 | 57 | 55
  Induration/Papulation - Trunk: -2 = Improve by 2 | 31 | 33 | 34
  Induration/Papulation - Trunk: -3 = Improve by 3 | 0 | 0 | 0
  Induration/Papulation - Upper Limbs: 3 = Worsen by 3 | 0 | 0 | 0
  Induration/Papulation - Upper Limbs: 2 = Worsen by 2 | 0 | 2 | 1
  Induration/Papulation - Upper Limbs: 1 = Worsen by 1 | 4 | 5 | 6
  Induration/Papulation - Upper Limbs: 0 = No change | 75 | 79 | 88
  Induration/Papulation - Upper Limbs: -1 = Improve by 1 | 83 | 83 | 81
  Induration/Papulation - Upper Limbs: -2 = Improve by 2 | 39 | 35 | 26
  Induration/Papulation - Upper Limbs: -3 = Improve by 3 | 0 | 1 | 1
  Induration/Papulation - Lower Limbs: 3 = Worsen by 3 | 0 | 0 | 0
  Induration/Papulation - Lower Limbs: 2 = Worsen by 2 | 0 | 1 | 1
  Induration/Papulation - Lower Limbs: 1 = Worsen by 1 | 5 | 2 | 6
  Induration/Papulation - Lower Limbs: 0 = No change | 100 | 100 | 116
  Induration/Papulation - Lower Limbs: -1 = Improve by 1 | 71 | 81 | 57
  Induration/Papulation - Lower Limbs: -2 = Improve by 2 | 24 | 21 | 23
  Induration/Papulation - Lower Limbs: -3 = Improve by 3 | 1 | 0 | 0
  Lichenification - Head & Neck: 3 = Worsen by 3 | 0 | 0 | 0
  Lichenification - Head & Neck: 2 = Worsen by 2 | 1 | 1 | 1
  Lichenification - Head & Neck: 1 = Worsen by 1 | 5 | 5 | 2
  Lichenification - Head & Neck: 0 = No change | 131 | 137 | 151
  Lichenification - Head & Neck: -1 = Improve by 1 | 47 | 41 | 42
  Lichenification - Head & Neck: -2 = Improve by 2 | 17 | 20 | 7
  Lichenification - Head & Neck: -3 = Improve by 3 | 0 | 1 | 0
  Lichenification - Trunk: 3 = Worsen by 3 | 0 | 0 | 0
  Lichenification - Trunk: 2 = Worsen by 2 | 0 | 0 | 1
  Lichenification - Trunk: 1 = Worsen by 1 | 4 | 6 | 6
  Lichenification - Trunk: 0 = No change | 114 | 126 | 127
  Lichenification - Trunk: -1 = Improve by 1 | 59 | 50 | 50
  Lichenification - Trunk: -2 = Improve by 2 | 24 | 23 | 17
  Lichenification - Trunk: -3 = Improve by 3 | 0 | 0 | 2
  Lichenification - Upper Limbs: 3 = Worsen by 3 | 0 | 0 | 0
  Lichenification - Upper Limbs: 2 = Worsen by 2 | 0 | 2 | 1
  Lichenification - Upper Limbs: 1 = Worsen by 1 | 7 | 6 | 12
  Lichenification - Upper Limbs: 0 = No change | 93 | 93 | 98
  Lichenification - Upper Limbs: -1 = Improve by 1 | 72 | 83 | 65
  Lichenification - Upper Limbs: -2 = Improve by 2 | 29 | 18 | 26
  Lichenification - Upper Limbs: -3 = Improve by 3 | 0 | 3 | 1
  Lichenification - Lower Limbs: 3 = Worsen by 3 | 0 | 0 | 0
  Lichenification - Lower Limbs: 2 = Worsen by 2 | 0 | 1 | 1
  Lichenification - Lower Limbs: 1 = Worsen by 1 | 6 | 2 | 5
  Lichenification - Lower Limbs: 0 = No change | 126 | 113 | 126
  Lichenification - Lower Limbs: -1 = Improve by 1 | 54 | 71 | 52
  Lichenification - Lower Limbs: -2 = Improve by 2 | 13 | 16 | 18
  Lichenification - Lower Limbs: -3 = Improve by 3 | 2 | 2 | 1
  Pruritus: 3 = Worsen by 3 | 0 | 1 | 0
  Pruritus: 2 = Worsen by 2 | 2 | 1 | 0
  Pruritus: 1 = Worsen by 1 | 4 | 5 | 10
  Pruritus: 0 = No change | 42 | 41 | 59
  Pruritus: -1 = Improve by 1 | 76 | 78 | 82
  Pruritus: -2 = Improve by 2 | 73 | 71 | 49
  Pruritus: -3 = Improve by 3 | 4 | 8 | 3

4. Secondary Outcome: Evaluation of Application Site Reactions
Description: Dryness, burning/stinging, erosion, edema, and pain
Time Frame: Day 15
Population: Safety with data for this parameter
Measure: Count of Participants; unit: Participants
Arm/Group | Test | Reference Standard | Placebo
Number analyzed (Participants) | 214 | 213 | 217
Participants
  Dryness: None | 121 | 126 | 103
  Dryness: Mild | 64 | 63 | 76
  Dryness: Moderate | 23 | 21 | 33
  Dryness: Severe | 6 | 3 | 5
  Stinging/Burning: None | 180 | 171 | 172
  Stinging/Burning: Mild | 23 | 30 | 28
  Stinging/Burning: Moderate | 11 | 11 | 14
  Stinging/Burning: Severe | 0 | 1 | 3
  Erosion: None | 190 | 187 | 190
  Erosion: Mild | 14 | 19 | 18
  Erosion: Moderate | 8 | 7 | 9
  Erosion: Severe | 2 | 0 | 0
  Edema: None | 196 | 194 | 193
  Edema: Mild | 14 | 13 | 17
  Edema: Moderate | 4 | 6 | 7
  Edema: Severe | 0 | 0 | 0
  Pain: None | 192 | 195 | 197
  Pain: Mild | 18 | 16 | 12
  Pain: Moderate | 4 | 2 | 7
  Pain: Severe | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 15
Description: Serious Adverse Event: substantial disruption of the ability to conduct normal functions was not included in the study protocol definition
Arm/Group | Test | Reference Standard | Placebo
All-Cause Mortality (participants affected / at risk) | 0/215 | 0/214 | 0/220
Serious Adverse Events (participants affected / at risk) | 0/215 | 0/214 | 0/220
Other Adverse Events (participants affected / at risk) | 0/215 | 0/214 | 0/220

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The publication rights for the data generated rests with the sponsor. The site retains the right to use such data or results for its own publication only upon getting the written approval from the sponsor, only after the first publication of such data by the sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-10-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT03107611/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/11/NCT03107611/SAP_001.pdf